CLINICAL TRIAL: NCT02316171
Title: A Phase 1 Study to Evaluate the Safety and Clinical Activity of Intravesicular CAVATAK (Coxsackievirus A21, CVA21) Alone and in Sequential Combination With Low Dose Mitomycin C in Patients With Non-Muscle Invasive Bladder Cancer (VLA-012 CANON)
Brief Title: CAVATAK (CVA21) in Non-muscle Invasive Bladder Cancer (VLA-012 CANON)
Acronym: CANON
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: V937-008; VLA-012 (Other: Viralytics Study ID); 2014-003938-81 (EudraCT Number)
Record Dates: First submitted 2014-12-07; First posted 2014-12-12 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: Coxsackievirus A21; bladder cancer; CVA21; CAVATAK
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVA21 (Experimental): CVA21 was administered by intravesical instillation at one of three (3) ascending dose levels or schedules.
  Interventions: Biological: CVA21
- CVA21/Mitomycin C (Experimental): Mitomycin C (MMC) was administered at 10 mg by intravesical instillation on Day 1. Four hours after instillation of MMC, CVA21 was administered by intravesical instillation of one of 2 ascending dose levels or schedules. Subjects received a second instillation of CVA21 alone on Day 2 without pretreatment with MMC.
  Interventions: Biological: CVA21; Drug: Mitomycin C

INTERVENTIONS:
Biological: CVA21 — CAVATAK is a purified preparation of CVA21
  Other Names: CAVATAK, Coxsackievirus A21
Drug: Mitomycin C — Chemotherapy
  Arms: CVA21/Mitomycin C

SUMMARY:
The study consisted of 2 sequential parts. Part A assessed the safety and tolerability of CAVATAK administered via intravesical instillation in patients with non-muscle invasive bladder cancer scheduled to undergo TUR. Part B assessed the safety and tolerability of CAVATAK administered in sequential combination with low dose Mitomycin C in the same patient population.

DETAILED DESCRIPTION:
This was a Phase I, two-part, open-label, dose-escalation study designed to evaluate CVA21 alone and in sequential combination with low-dose mitomycin C in patients with non-muscle invasive bladder cancer (NMIBC) who were candidates for and were planning to undergo TUR for treatment of their disease. This gave a relatively homogeneous study population and facilitated collection of resected tumour tissue for histological, pharmacodynamics (PD) and pharmacokinetic (PK) analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NMIBC based on cystoscopic appearance
* ECOG 0-2
* No intravesical therapy within 6 weeks of study entry
* No prior radiation to the pelvis
* ANC >1500/mm³; Hb >9.0 g/dL; Platelet >100000/mm³
* Serum creatinine ≤ 1.5 mg/dL
* Bilirubin within normal limits; AST ≤ 2.5x upper limit of normal (ULN); ALT ≤ 2.5 x ULN; alkaline phosphatase ≤ 2.5x ULN unless bone metastasis is present in the absence of liver metastasis
* INR < 1.2; aPPT = 0.8-1.2; PT = 0.9-1.8
* Candidate for TUR and planning to undergo TUR
* Negative pregnancy test within 7 days of treatment start
* Patients of child-bearing potential must agree to use an effective method of birth control

Exclusion Criteria:

* Prior local or systemic treatments for NMIBC
* Concurrent treatment with any chemotherapeutic agent
* Patients not deemed acceptable for general anaesthesia
* Women who are pregnant or lactating
* History of vesicoureteric reflux or an indwelling urinary stent
* Administration of an investigational agent within 3 months of study entry
* Active cardiac disease
* Known infection with HIV, hepatitis B or C
* Active uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2016-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hardev Pandha, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (1):
- University of Surrey, Guildford, United Kingdom

REFERENCES:
- [Result] Annels NE, Mansfield D, Arif M, Ballesteros-Merino C, Simpson GR, Denyer M, Sandhu SS, Melcher AA, Harrington KJ, Davies B, Au G, Grose M, Bagwan I, Fox B, Vile R, Mostafid H, Shafren D, Pandha HS. Phase I Trial of an ICAM-1-Targeted Immunotherapeutic-Coxsackievirus A21 (CVA21) as an Oncolytic Agent Against Non Muscle-Invasive Bladder Cancer. Clin Cancer Res. 2019 Oct 1;25(19):5818-5831. doi: 10.1158/1078-0432.CCR-18-4022. Epub 2019 Jul 4. PMID 31273010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 patients were enrolled into VLA012A and 6 patients into VLA012B and data presented for these 15 patients. One patient was enrolled, but not treated due to difficulties in placing the urinary catheter.
Groups:
- A1 - CVA21 1x10^8 TCID50: CAVATAK was administered by intravesical instillation at 1x10^8 TCID50.
- A2 - CVA21 3x10^8 TCID50.: CAVATAK was administered at 3x10^8 TCID50
- A3 - CVA21 3x10^8 TCID50 x2: CAVATAK was administered at 3x10^8 TCID50 twice.
Period: Overall Study
Arm/Group | A1 - CVA21 1x10^8 TCID50 | CVA21/Mitomycin C | A2 - CVA21 3x10^8 TCID50. | A3 - CVA21 3x10^8 TCID50 x2
Started | 4 | 6 | 3 | 3
Completed | 3 | 6 | 3 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — difficulties with urinary catheter | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Received at least one dose of treatment.
Groups:
- CVA21: CVA21 was administered by intravesical instillation of one of 3 ascending dose levels or schedules:
- CVA21/MitomycinC: Mitomycin C (MMC) was administered at 10 mg by intravesical instillation on Day 1. Four hours after instillation of MMC, CVA21 was administered by intravesical instillation of one of 2 ascending dose levels or schedules. Subjects received a second instillation of CVA21 alone on Day 2 without pretreatment with MMC
- Total: Total of all reporting groups
Arm/Group | CVA21 | CVA21/MitomycinC | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11.6) | 62.7 (8.3) | 65 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicities Treatment-related Adverse Events.
Description: Number of Participants with Treatment-emergent adverse events. The events for each cohort of dose of CVA21 only are pooled for the analysis.
Time Frame: 30 days from last dose
Measure: Count of Participants; unit: Participants
Groups:
- CVA21: CVA21 was administered by intravesical instillation of one of 3 ascending dose levels or schedules
Arm/Group | CVA21 | CVA21/Mitomycin C
Number analyzed (Participants) | 9 | 6
Participants | 9 | 6

ADVERSE EVENTS:
Time Frame: 30 days. The analysis for each dose escalation cohort for CVA21 only was pooled as the numbers were so small. This resulted in an analysis showing 2 arms.
Description: No SUSARs were reported for the VLA-012 study.
Arm/Group | CVA21 | CVA21/Mitomycin C
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/6
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVA21 (N=9) | CVA21/Mitomycin C (N=6)
E. Coli urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVA21 (N=9) | CVA21/Mitomycin C (N=6)
Hematuria (Renal and urinary disorders) | 5 (5) | 4 (4)
Dysuria (Renal and urinary disorders) | 5 (5) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 2 (2) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 0 (0)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) — General disorders and administration site conditions
Chills (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Influenza like illness (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Pyrexia (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Genital discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects with limited follow-up; study not designed to give any indication of efficacy. The analysis for each dose escalation cohort for CVA21 only was pooled as the numbers were so small. This resulted in an analysis showing 2 arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes